CLINICAL TRIAL: NCT00895102
Title: An Open-Label Randomized, Crossover Study to Evaluate the Bioavailability of ABT-333 Tablets Versus Capsules, and A Double-blind, Randomized, Crossover Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profiles of Single Ascending Doses of ABT-333 Tablets Versus Placebo in Healthy Volunteers
Brief Title: Bioavailability of ABT-333 Tablet Versus First in Human (FIH) Capsule Formulation and Safety, Tolerability and PK Study of Single Doses of ABT-333 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Daniel Cohen, MD/Study Medical Director, Abbott
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: M11-032
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-09

CONDITIONS: HCV Infection
Keywords: Bioavailability (BA); Single Ascending Dose (SAD)
MeSH Terms: conditions — Hepatitis C | interventions — dasabuvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. ABT-333 Capsule vs ABT-333 Tablet (Active Comparator): 400mg ABT-333 Tablet, QD, single dose vs eight 50mg ABT-333 Capsules, QD, single dose
  Interventions: Drug: ABT-333 Tablet; Drug: ABT-333 Capsule
- 2. ABT-333 Tablet (Active Comparator): ABT-333 400mg Tablet, QD, single ascending doses (1200mg, 1600mg, 2400mg)
  Interventions: Drug: ABT-333 Tablet; Drug: Placebo
- 3. Placebo (Placebo Comparator): Placebo tablets, QD, single ascending doses
  Interventions: Drug: ABT-333 Tablet; Drug: Placebo

INTERVENTIONS:
Drug: ABT-333 Tablet — See Arm Description for more information.
  Other Names: ABT-333
Drug: Placebo — See Arm Description for more information.
  Arms: 2. ABT-333 Tablet; 3. Placebo
Drug: ABT-333 Capsule — See arm description for more information
  Arms: 1. ABT-333 Capsule vs ABT-333 Tablet

SUMMARY:
The purpose of this study is to determine the bioavailability, pharmacokinetic and safety profiles of an experimental Hepatitis C virus (HCV) polymerase inhibitor in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* overall healthy subjects;
* non-childbearing potential females included

Exclusion Criteria:

* history of significant sensitivity to any drug;
* positive test for HAV IgM, HBsAg, anti-HCV Ab or anti-HIV Ab;
* history of gastrointestinal issues or procedures;
* history of seizures, diabetes or cancer (except basal cell carcinoma);
* clinically significant cardiovascular, respiratory (except mild asthma), renal, gastrointestinal, hematologic, neurologic, thyroid, or any uncontrolled medical illness or psychiatric disorder;
* use of tobacco or nicotine-containing products with the 6-month period prior to study drug administration;
* donation or loss of 550 mL or more blood volume or receipt of a transfusion of any blood product within 8 weeks prior to study drug administration;
* abnormal screening laboratory results that are considered clinically significant by the investigator;
* current enrollment in another clinical study;
* previous enrollment in this study;
* recent (6-month) history of drug/alcohol abuse that could preclude adherence to the protocol;
* pregnant or breastfeeding female;
* requirement for any OTC and/or prescription medication, vitamins and/or herbal supplements on a regular basis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine relative bioavailability of the ABT-333 tablet formulation compared to the FIH capsule formulation | 2 days post dosing
To evaluate single dose safety and tolerability of a ABT-333 tablet formulation relative to placebo | 2 days post dosing
To evaluate single dose pharmacokinetics of a ABT-333 tablet formulation | 2 days post dosing
Pharmacokinetics | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cohen, MD, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 19441, Waukegan, Illinois, United States